CLINICAL TRIAL: NCT04346121
Title: Non-COVID Patient-safety Incidents Reported by General Practitioners in Time of Lockdown: Protocol for a Cross-sectional Descriptive Study.
Brief Title: Non-COVID Patient-safety Incidents Reported by General Practitioners in Time of Lockdown: Protocol for a Cross-sectional Descriptive Study.cRisis
Acronym: PSI-RECORd-GP
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0182
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Patient Safety
Keywords: Safety care, COVID, primary care, organization of care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: GPs reports of potential patient safety incidents, non-COVID-19 related — GPs reports of potential patient safety incidents, non-COVID-19 related

SUMMARY:
The COVID-19 epidemic is causing a global health crisis. In France, it has imposed a major reorganization of the healthcare system. This emergency reorganization is unprecedented. It involved first, second and third line care. Following this reorganization and from the first days of confinement, a decrease in care activity not related to COVID-19 was observed in médical offices, in emergency services, and in secondary and tertiary care services. This decrease in activity could indicate a decrease in pathologies related to work, transportation or non-COVID-19 infections, due to a favourable effect of lockdown. Nevertheless, some health professionals report the opposite in the media and on social networks, an unusual increase in events (appendicular peritonitis treated late, increase in domestic violence, etc.), while others are surprised by a decrease in activity that is difficult to explain (leukaemia diagnoses by biologists, for example). One hypothesis is that such changes could be related to the reorganisation of the health care system or to the consequences of lockdown.

The World Health Organization (WHO) recommends a systematic collection and analysis of patient safety incidents (also called "adverse events" in France). The objective is to assess the roles of the system and human factors in patient safety, in order to propose changes to the global system and local organisation. In France, there is a system for reporting serious adverse events related to care. Only 4% of the 820 serious adverse events reported in 2018 were reported by primary healthcare professionals (1). However, patient safety incidents in primary care are known to have specific mechanisms, types and mechanisms (2).

We hypothesize that the COVID-19 health crisis may have induced unusual patient safety incidents through new mechanisms in a context associating reorganization of the healthcare system and population lockdown. Such a scenario requires the implementation of a massive collection of potential incidents and their systematic and well-structured analysis.

Thus, the objective of our study is to describe patient safety incidents related to the reorganization of care and/or lockdown in the context of the COVID-19 health crisis (types, severity, mechanisms) reported by general practitioners in France.

1. HAS. Retour d'expérience sur les événements indésirables graves associés à des soins (EIGS) [Internet]. [cited 2020 Apr 7]. Available from: https://www.has-sante.fr/jcms/c_2882289/fr/retour-d-experience-sur-les-evenements-indesirables-graves-associes-a-des-soins-eigs
2. Carson-Stevens A, Hibbert P, Avery A, Butlin A, Carter B, Cooper A, et al. A cross-sectional mixed methods study protocol to generate learning from patient safety incidents reported from general practice. BMJ Open. 2015 Dec 1;5(12):e009079.

ELIGIBILITY:
Inclusion Criteria:

* General practitioners practising in primary care, in France, who have given their consent to receive e-mails from the Collège National des Généralistes Enseignants (CNGE)
* Any patient undergoing primary care

Exclusion Criteria:

* Other primary health care professionals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General practitioners will be invited via an email issued to report potential patient safety incidents unrelated to COVID-19 that they have observed since March 14, 2020 (date of entry into Stage 3 of the COVID-19 epidemic)
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Describe patient safety incidents (types, severity, contributing and correcting factors) - 1000 PSI required | 6 months
  Describe patient safety incidents (types, severity, contributing and correcting factors) by the reorganization of care and/or lockdown reported by French GPs in the context of the COVID-19 health crisis - 1000 PSI required
Describe patient safety incidents (types, severity, contributing and correcting factors) - 100 PSI required | 2 months
  Describe patient safety incidents (types, severity, contributing and correcting factors) by the reorganization of care and/or lockdown reported by French GPs in the context of the COVID-19 health crisis - 100 PSI required

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal FOURNIER, Doctor, Study Chair — Nantes University Hospital
Locations (1):
- University Hospital, Nantes, France

REFERENCES:
- [Derived] Fournier JP, Amelineau JB, Hild S, Nguyen-Soenen J, Daviot A, Simonneau B, Bowie P, Donaldson L, Carson-Stevens A. Patient-safety incidents during COVID-19 health crisis in France: An exploratory sequential multi-method study in primary care. Eur J Gen Pract. 2021 Dec;27(1):142-151. doi: 10.1080/13814788.2021.1945029. PMID 34212814